CLINICAL TRIAL: NCT01385540
Title: Exploration of Cortical Neural Network in Patients With Bothersome Tinnitus
Status: Terminated | Type: Observational
Why Stopped: Study tasks to difficult for subjects to complete.
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Tinnitus Association (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine, Washington University School of Medicine
Other Study IDs: 201106289
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Tinnitus
Keywords: Tinnitus, fMRI, task-based fMRI, attention network
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Task-based fMRI
  Interventions: Behavioral: Task-Based Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Behavioral: Task-Based Functional Magnetic Resonance Imaging (fMRI) — Individuals will be shown a target, which is randomly selected from 12 objects designated as targets, before each scan. The target for a scan will never appear as a non-target object in another scan. Per established protocol, individuals will fixate on a central cross prior to imaging. Individuals will press a MR-compatible button when they detect the target. Target objects only appear in the cued stream. Cues, a filled red square, are programmed to occur, on average, every 2.06, 4.12, or 6.18 seconds within a temporal window of ± 400 milliseconds centered on those values.

SUMMARY:
This will be an experimental task-based functional MRI pilot study involving the neuroimaging assessment of patients with severely bothersome tinnitus, defined by a global bothersome scale. The investigators plan to enroll a total of 12 participants (6 severely bothered tinnitus and 6 age-matched non-tinnitus controls) over the course of six months to undergo task-based imaging. Subjects in the tinnitus group may have previously participated in the CTRWU study (HRPO: 07-0689) conducted by Dr. Jay Piccirillo at Washington University and have given permission to be contacted for consideration in future studies. The selected paradigm will allow us to advance knowledge about the role of the attention, control, and other cortical networks in the development and maintenance of bothersome tinnitus.

DETAILED DESCRIPTION:
Task-Based Functional Magnetic Resonance Imaging (fMRI) The task-based fMRI protocol is based on work performed at Washington University by Dr. Gordon Shulman and published in The Journal of Neuroscience.(Shulman, Astafiev, Franke, Pope, Snyder, McAvoy, and Corbetta 2009) Individuals will be shown a target, which is randomly selected from 12 objects designated as targets, before each scan. The target for a scan will never appear as a non-target object in another scan. Per established protocol, individuals will fixate on a central cross prior to imaging. Individuals will press a MR-compatible button when they detect the target. Target objects only appear in the cued stream. Cues, a filled red square, are programmed to occur, on average, every 2.06, 4.12, or 6.18 seconds within a temporal window of ± 400 milliseconds centered on those values.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 to 60 years
* Subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or greater
* Either "moderately bothered" or "severely bothered" on the Global Bothersome scale
* THI score of ≥ 30.
* Able to give written informed consent
* Able to read, write, speak and understand English fluently

Exclusion Criteria:

* Tinnitus related to cochlear implantation, retrocochlear lesion, or other known anatomic lesions of the ear and temporal bone
* History of Ménière's Disease
* History of hyperacusis or misophonia (hyper-sensitivity to noises)
* Cardiac pacemakers, intracardiac lines, implanted medication pumps, implanted electrodes in the brain, or any other contraindication for MRI scan
* An acute or chronic unstable medical condition which, in the opinion of the investigator, would require stabilization prior to testing.
* Any active ear disease that, in the opinion of the PI or mentor, needs to be further evaluated
* A Short Blessed Test score of 9 or greater
* PHQ-9 score ≥ 10; consistent with diagnosis of moderate depression.
* History of seizure disorder or other neurological condition.
* Any psychiatric co-morbidity that may complicate the interpretation of study results. Subjects may not be currently taking antidepressants.
* Any tinnitus related to a Workman's Compensation claim or litigation-related event
* Currently pregnant: Women of childbearing potential must have a negative urine pregnancy test prior to MRI
* Weight over 300 pounds
* History of claustrophobia
* Inability to lay flat for 2 hours
* Active alcohol and/or drug dependence or history of alcohol and/or drug dependence within the last year
* Any medical condition that, in the opinion of the investigators, confounds study results or places the subject at greater risk
* Unable to provide written informed consent
* Blindness or inability to see screen for task-based testing without eyeglasses, subjects may wear contacts if able to lie flat and keep eyes focused on testing screen for up to 2 hours.
* Previous participation in a task-based MRI study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Target population will consist of 12 adult participants - 6 with moderately, severely or worse, bothersome tinnitus, based on both a global bothersome score (i.e. How bothered are you by your tinnitus?) and the Tinnitus Handicap Index (THI). THI is a 25-question survey designed to assess how much tinnitus affects a person-possible scores range from 0-100, with a score 38 falling in the 75th percentile. The other six participants (Control group) will be age-matched without tinnitus.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States